CLINICAL TRIAL: NCT03213626
Title: A Phase II Trial of Cabozantinib and Erlotinib for Patients With EGFR and c-Met Co-expressing Metastatic Pancreatic Adenocarcinoma
Brief Title: Cabozantinib and Erlotinib for Patients With EGFR and c-Met Co-expressing Metastatic Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There were no objective responses by patient 7.
Sponsor: Patrick Joseph Loehrer Sr. (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Patrick Joseph Loehrer Sr., Associate Dean for Cancer Research Director, Indiana University Melvin and Bren Simon Cancer Center, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0597
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — cabozantinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib + erlotinib (Experimental)
  Interventions: Drug: Cabozantinib 40 MG; Drug: Erlotinib 100Mg Tab

INTERVENTIONS:
Drug: Cabozantinib 40 MG — To be taken orally once daily
Drug: Erlotinib 100Mg Tab — To be taken orally once daily

SUMMARY:
This is an open-label, single arm, phase II trial. Safety will be monitored on an ongoing basis. Laboratory testing (chemistry, hematology tests) will be performed every 2 weeks for the first 8 weeks followed by assessments every 4 weeks. Other safety evaluations including EKGs, urinalysis, coagulation and thyroid function studies will be performed at regular intervals.

Adverse event seriousness, severity grade, and relationship to study treatment will be assessed by the investigator. Severity grade will be defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

Tumors will be assessed by contrast enhanced CT or MRI every 8 weeks. Pre-treatment tissue will be obtained via CT-guided FNA biopsy or collected during resection. However, archival tissue will also be requested, when available and if adequate for testing. Post-treatment tissue will be obtained on Day 15 (i.e., Week 3/Day 1) via CT-guided FNA biopsy. All tumor tissue from eligible patients will be utilized for the correlative studies which are outlined in this trial.

Each subject's course will consist of three periods:

* A Pre-Treatment Period in which subjects are consented and undergo screening assessments to be qualified for the study;
* A Treatment Period in which subjects receive study treatment and undergo study assessments. Patients who meet the eligibility criteria will be treated with cabozantinib orally at 40 mg daily and erlotinib orally at 100 mg daily without breaks;
* A Post-Treatment Period in which subjects no longer receive study treatment but undergo follow-up study assessments and contacts.

DETAILED DESCRIPTION:
Primary Objective The primary objective of this trial is to demonstrate a radiographic response rate of 15% or greater for the combination in a selected population.

Secondary Objectives

The secondary objectives of this trial are:

* To estimate progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), overall survival (OS); and
* To assess safety and tolerability of this combination in the target patient population.

Correlative Objectives

The following tests will be performed on blood and tumor tissue samples collected during this trial to correlate with PFS and OS:

* c-Met and EGFR mRNA by RT-qPCR
* plasma HGF and soluble Met receptor
* c-Met and EGFR phosphoprotein levels by IHC
* KRAS mutation status

ELIGIBILITY:
Inclusion Criteria

A subject must fully meet all of the following criteria to be eligible for the study:

1. The subject has a biopsy-proven diagnosis of adenocarcinoma of the pancreas (or recurrence of previously resected disease) with metastatic disease that is measurable per RECIST 1.1;
2. The subject must have tumor that is amenable to fine needle biopsy via computerized tomography (CT) guided approach OR an archived tissue sample such as a prior surgical sample or biopsy sample that is adequate for testing;
3. The subject must have EGFR and c-Met overexpressed in tumor as determined by immunohistochemistry (IHC) test score of 2+ for both markers;
4. The subject has demonstrated radiographic progression after front-line treatment for locally advanced or metastatic disease (prior adjuvant therapy allowed if ≥ 6 months elapsed between end of adjuvant therapy and metastatic relapse);
5. The subject is ≥ 18 years old on the day of consent;
6. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. The subject has recovery to baseline or ≤ Grade 1 CTCAE v.4.03 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy;
8. The subject has organ and marrow function and laboratory values as follows within 7 days before the first dose of study treatment:

   1. The ANC ≥ 1500/mm3 without colony stimulating factor support;
   2. Platelets ≥ 100,000/mm3;
   3. Hemoglobin ≥ 9 g/dL;
   4. Bilirubin ≤ 1.5 x the ULN. For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL;
   5. AST/ALT ≤ 3 x the ULN;
   6. Serum albumin ≥ 2.8 g/dl;
   7. Serum creatinine ≤ 1.5 x the ULN or creatinine clearance (CrCl) ≥ 40 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

   i. Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72); ii. Female: Multiply above result by 0.85; h. UPCR ≤ 1; i. Serum phosphorus, calcium, magnesium and potassium ≥ LLN; j. Prothrombin time (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x the ULN within 7 days before the first dose of study treatment;
9. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document;
10. The subject has a life expectancy of 12 weeks or greater;
11. The subject is able to tolerate oral medications and no evidence of ongoing malabsorption;
12. All sexually active subjects of reproductive potential must agree to use both a medically accepted barrier method (e.g., male or female condom) and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s);
13. Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy or bilateral oophorectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

1. The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment;
2. Prior treatment with cabozantinib or erlotinib;
3. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible;
4. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment;
5. The subject has received any other type of investigational agent within 28 days before the first dose of study treatment;
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment;
7. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel); Note: Low-dose aspirin for cardioprotection (per local applicable guidelines) and low-dose LMWH are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
8. The subject has experienced any of the following:

   1. clinically-significant GI bleeding within 6 months before the first dose of study treatment;
   2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment;
   3. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment; and
   4. clinically confirmed history of interstitial lung disease (ILD).
9. The subject has radiographic evidence of cavitating pulmonary lesion(s);
10. The subject has tumor invading or encasing any major blood vessels;
11. The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib;
12. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    a. Cardiovascular disorders including: i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening; ii. Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment; iii. Any history of congenital long QT syndrome; iv. Any of the following within 6 months before the first dose of study treatment:
    * unstable angina pectoris;
    * clinically-significant cardiac arrhythmias;
    * stroke (including transient ischemic attack (TIA), or other ischemic event);
    * myocardial infarction. b. GI disorders particularly those associated with a high risk of perforation or fistula formation including: i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before first dose of study treatment Note: Complete healing of an intra-abdominal abscess must be confirmed prior first dose of study treatment c. Other clinically significant disorders that would preclude safe study participation;
13. Major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible;
14. QTcF > 500 msec within 1 month before the first dose of study treatment:

    a. Three ECGs must be performed for eligibility determination. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
15. Pregnant or lactating females;
16. Active smoker;
17. Inability to swallow intact tablets;
18. Previously identified allergy or hypersensitivity to components of the study treatment formulations;
19. Diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy; malignancy felt by investigator to potentially affect subject survival or ability to evaluate disease response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single arm two stage design. The 1st stage was to have 11 patients and be terminated if 0 responded. The 2nd stage would have a total of 37 patients and if the number responding was <= 2, the combination was to be rejected. The study was terminated prematurely due to no patient benefit at Patient 7.
Period: Overall Study
Arm/Group | Cabozantinib + Erlotinib
Started | 7
Completed | 0
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 1
ECOG Performance Status [Count of Participants; unit: Participants]
  0-Fully active | 4
  1-Restricted in physically strenuous activity | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective (Radiographic) Response
Description: Percent of patients with Objective response and the Binomial Exact 95% confidence interval. Objective response is defined as having a best response of Complete Response (defined as disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10mm) or Partial Response (defined as at least a 30% decrease in the sum of diameters of target lesions from the baseline sum diameters) by RECIST v1.1 criteria.
Time Frame: 8 weeks
Population: All patients who received at least one dose of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
percentage of participants | 0

2. Secondary Outcome: Disease Control Rate
Description: Percent of patients achieving disease control and the Binomial Exact 95% confidence interval. Disease control is defined as having a best response of Complete Response (defined as disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10mm) or Partial Response (defined as at least a 30% decrease in the sum of diameters of target lesions from the baseline sum diameters) or Stable Disease for at least 4 months (defined by neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progression) by RECIST v1.1 criteria.
Time Frame: 8 weeks
Population: All patients who received at least one dose of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
percentage of participants | 0 [NA to NA] — There were no patients achieving disease control rate and the confidence interval was not calculated.

3. Secondary Outcome: Progression Free Survival
Description: Duration of time from the start of treatment to time of documented progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients who do not progress or die will be censored on their last evaluation date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: 2 years
Population: All patients who received at least one dose of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
months | 1.8 [0.7 to 1.9]

4. Secondary Outcome: Overall Survival
Description: Duration of time from the start of treatment to time of death due to any causes. Patients who do not die will be censored on their last known alive date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: 2 years
Population: All patients who received at least one dose of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
months | 7.7 [2.1 to 12.0]

5. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse events with grade >= 3.
Time Frame: Up to 5 months
Population: All patients who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib + Erlotinib
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 5 months for Adverse Events (Serious and Other). Up to 2 years for All Cause Mortality.
Arm/Group | Cabozantinib + Erlotinib
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib + Erlotinib (N=7)
Small intestinal obstruction (Gastrointestinal disorders) | 1
Biliary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib + Erlotinib (N=7)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT03213626/Prot_SAP_000.pdf